CLINICAL TRIAL: NCT00501735
Title: Single Agent Phase II Study of Forodesine (BCX1777) in the Treatment of Cutaneous T-Cell Lymphoma
Brief Title: Forodesine in the Treatment of Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-203
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Cutaneous T-cell Lymphoma (CTCL),
Keywords: T-Cell; Lymphoma; Forodesine; Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma; Mycosis Fungoides | interventions — forodesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Forodesine 200 mg — 2 x 100mg tablets once daily

SUMMARY:
This is a Phase II, non-randomized, open-label, single-arm trial that will be conducted at up to 50 sites in North America, Europe and Australia. This study is designed to assess objective response (OR) [complete response (CR) or partial response (PR)] in subjects with cutaneous manifestations of CTCL with a requirement for maintenance of such objective response for at least 28 days in subjects with stage IIB, III, and IVA CTCL. Additionally, this study will evaluate the safety and tolerability of CTCL subjects Stages IB, IIA, IIB, III, or IVA treated with oral forodesine.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females aged ≥18 years;
* Histologically confirmed diagnosis of CTCL, including mycosis fungoides and/or Sezary syndrome, documentation of diagnosis by histologic examination should be available;
* Subjects with CTCL stages IB, IIA, IIB, III, or IVA at the screening visit (i.e. stage refers to stage at study entry) and who have persistent, progressive, or recurrent disease during or following treatment with at least three forms of systemic therapy, one of which must have been oral bexarotene, unless treatment with oral bexarotene was not tolerated or was medically contraindicated;
* Anticipated life expectancy greater than 6 months;
* Performance status of 0, 1, or 2 by Eastern Cooperative Oncology Group (ECOG) criteria;
* Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of study treatment;
* Females of childbearing potential and sexually active males, if indicated, must be willing and able to use method(s) of contraception that are adequate to prevent or minimize the risk of pregnancy for the duration of the study;
* Written informed consent to participate in the study.

Exclusion Criteria:

* Proven or suspected extracutaneous visceral CTCL involvement (M1) (CTCL stage IVB) (note: presence of lymphadenopathy is permitted);
* Previous treatment with Forodesine;
* ECOG performance status >2;
* Concomitant use of any anti-cancer therapy or immune modifier;
* Concomitant use of any investigational agent or device;
* Concurrent treatment with any other anti-CTCL therapy, or radiation therapy [topical corticosteroids (classes 1 and 2 prohibited) or low dose oral corticosteroids (≤10 mg/day prednisone or equivalent) will not be excluded, but if used, must be a stable dose and schedule during the four weeks immediately prior to study entry];
* Use of previous therapies for CTCL within the timeframes specified below:

  1. Phototherapy in the previous 30 days;
  2. Electron beam therapy, photopheresis, systemic anticancer therapy, interferon therapy, or other investigational therapy in the previous 30 days;
  3. Oral retinoid (including bexarotene) in the previous 30 days
  4. Alemtuzumab (Campath) or other monoclonal antibody within the previous 30 days
  5. Vorinostat or other HDAC inhibitor within previous 30 days
  6. Any investigational therapy within the previous 30 days;
* ALT or AST >3 times ULN or alkaline phosphatase >2 times ULN;
* Calculated creatinine clearance ≤50 mL/min or serum creatinine ≥1.8 mg/dL;
* Serum potassium <3.3 mg/dL or >5.5 mg/dL;
* Evidence of clinically significant (uncontrolled) hypo- or hyperthyroidism;
* Recent (in past 6 months) medically significant cardiac event (i.e., myocardial infarction, cardiac surgery);
* Presence of congestive heart failure (NYHA class IV) or angina (NYHA class IV) or presence of a medically significant dysrhythmia;
* Presence of any of the following ECG findings:

  1. Congenital long QT syndrome;
  2. QTc interval >480 msec (Bazett's correction);
* Presence of uncontrolled hypertension manifested by systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥90 mmHg;
* Hemoglobin <9.0 gm/dL (intermittent red blood cell transfusions permitted);
* Absolute neutrophil count <1500 cells/mm3;
* Platelet count <75,000/mm3;
* Requirement for neutrophil or platelet growth factor therapy or administration of such therapy in the previous 30 days;
* CD4 count <200/mm3;
* Documented current active infection with HIV, Hepatitis B, Hepatitis C, and/or CMV;
* Presence of uncontrolled bacterial or viral infection (subject may be receiving chronic antimicrobial therapy); or,
* History of culture-documented bacteremia in the previous 2 weeks;
* Recent (i.e., in past 2 weeks) change in doses or regimens of medications used for any chronic non-oncologic condition for reasons of worsening of the chronic illness (change in doses of chronic medications associated with improvement in a chronic illness are not exclusionary);
* Presence of any acute or chronic non-oncologic disease which, in the opinion of the investigator, is medically uncontrolled;
* Coexistent second malignancy or history of prior malignancy within previous 5 years [excluding basal cell or squamous cell carcinoma of skin and cervical neoplasia (carcinoma-in-situ) that has been treated curatively]. Surgically resected nonmelanomatous skin cancer (non-CTCL) with no evidence of recurrence in previous 6 months is permitted; and,
* Any significant medical or psychiatric condition that, in the opinion of the investigator, might prevent the subject from complying with all required study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the objective response rate to treatment with oral forodesine in subjects with cutaneous manifestations of CTCL subjects, stages IIB, III, and IVA. | Duration of Study

SECONDARY OUTCOMES:
Safety and tolerability | Duration of Study
Time to and duration of objective response in cutaneous manifestations | Duration of Study
Time to loss of objective response | Duration of Study
Objective response rate, time to and duration of extracutaneous manifestations | Duration of Study
Health related quality of life | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Nashat Gabrail, MD, Principal Investigator — Gabrail Cancer Center; Madeleine Duvic, MD, Principal Investigator — M.D. Anderson Cancer Center - Dermatology; Youn Kim, MD, Principal Investigator — Stanford University; Andres Forero-Torres, M.D., Principal Investigator — University of Alabama at Birmingham, Comprehensive Cancer Ctr.; Alan B Fleischer, Jr., MD, Principal Investigator — Wake Forest University Health Sciences; Gary S. Wood, MD, Principal Investigator — University of Wisconsin-Madison, Dept of Dermatology; Andre Goy, MD, Principal Investigator — Hackensack Universeity Medical Ctr; Larisa Geskin, MD, Principal Investigator — Hillman Cancer Ctr., University of Pittsburgh; Nancy Bartlett, MD, Principal Investigator — Washington University School of Medicine; Francine Foss, MD, Principal Investigator — Yale University; Miles Prince, MD, Principal Investigator — Cabrini Hospital; Elise Olsen, MD, Principal Investigator — Duke University; Sareeta S Parker, MD, Principal Investigator — Emory University; Neil J Korman, MD, PhD, Principal Investigator — University Hospitals Case Medical Ctr., Dept. of Dermatology; Francesco Turturro, MD, Principal Investigator — LSU Health Sciences Ctr., Feist-Weiller Cancer Center; Andrei R Shustov, MD, Principal Investigator — Seattle Cancer Care Alliance
Locations (41):
- United States (19):
  - University of Alabama at Birmingham, Comprehensive Cancer Ctr, Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - LSU Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Ctr, Hackensack, New Jersey
  - Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sceinces, Dept. of Dermatology, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals Case Medical Center, Dept. of Dermatology, Cleveland, Ohio
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Ctr., University of Pittsburgh, Pittsburgh, Pennsylvania
  - M.D. Anderson Cancer Center - Dermatology, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin-Madison, Dept of Dermatology, Madison, Wisconsin
- Cabrini Hospital, Malvern, Victoria, Australia
- Wien, Vienna, Austria
- Helsinki, Helsinki, Finland
- France (6):
  - Hopital Hotel-Dieu, Clermont-Ferrand
  - Creteil, Créteil
  - Montpellier, Montpellier
  - Pessac, Pessac
  - CHU Robert Debre, Reims
  - Toulouse, Toulouse
- Germany (4):
  - Campus Charité Mitte, Berlin
  - Universitatsklinikum Jena, Jena
  - Universitat Kiel, Kiel
  - Klinik fur Dermatologie, Venerologie und Allergologie, Mannheim
- Italy (5):
  - Bologna, Bologna
  - Firenze, Florence
  - Milan, Milan
  - Rome, Rome
  - Torino, Torino
- Madrid, Madrid, Spain
- Zurich, Zurich, Switzerland
- United Kingdom (2):
  - London, London
  - Manchester, Manchester

REFERENCES:
- [Derived] Dummer R, Duvic M, Scarisbrick J, Olsen EA, Rozati S, Eggmann N, Goldinger SM, Hutchinson K, Geskin L, Illidge TM, Giuliano E, Elder J, Kim YH. Final results of a multicenter phase II study of the purine nucleoside phosphorylase (PNP) inhibitor forodesine in patients with advanced cutaneous T-cell lymphomas (CTCL) (Mycosis fungoides and Sezary syndrome). Ann Oncol. 2014 Sep;25(9):1807-1812. doi: 10.1093/annonc/mdu231. Epub 2014 Jun 19. PMID 24948692